CLINICAL TRIAL: NCT02628886
Title: A Randomized, Controlled, Double-blind, Phase 3 Trial to Evaluate the Effects of Maternal or Neonatal Pneumococcal Conjugate Vaccination on Pneumococcal Carriage in Infants up to Nine Months of Age - The PROPEL Trial
Brief Title: Protecting From Pneumococcus in Early Life (The PROPEL Trial)
Acronym: PROPEL
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: WHO Pneumococcal Serology Reference Laboratory Institute of Child Health (Unknown); BUGS Bioscience London Bioscience Innovation Centre 2 Royal College Street London (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SCC 1433
Record Dates: First submitted 2015-12-07; First posted 2015-12-11 (Estimated); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Pneumonia
Keywords: maternal and neonatal pneumococcal conjugate vaccination; pneumococcal carriage
MeSH Terms: conditions — Pneumonia | interventions — 13-valent pneumococcal vaccine; Sodium Chloride; Tetanus Toxoid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- maternal group (Experimental): 13-valent pneumococcal conjugate vaccine [Prevenar13®] (PCV13) vaccine, 0.5ml, once, stat, plus tetanus toxoid to pregnant women between 28-34 weeks and their infants will get PCV13 at 8, 12 and 16 weeks according to normal EPI vaccination in country
  Interventions: Biological: 13-valent pneumococcal conjugate vaccine [Prevenar13®] plus tetanus toxoid
- control group (Placebo Comparator): placebo sterile 0.9% sodium chloride, 0.5ml, once, stat plus tetanus toxoid to pregnant women between 28-34 weeks and their infants will get PCV13 at 8, 12 and 16 weeks according to normal EPI vaccination in country
  Interventions: Biological: placebo 0.9% sodium chloride plus tetanus toxoid
- neonatal group (Experimental): tetanus toxoid to pregnant women between 28-34 weeks and their infants will get PCV 13 0.5ml at birth, 8 weeks and 16 weeks
  Interventions: Other: tetanus toxoid

INTERVENTIONS:
Biological: 13-valent pneumococcal conjugate vaccine [Prevenar13®] plus tetanus toxoid — pregnant women will be given intramuscular PCV 13 vaccine between 28-34 weeks
  Other Names: PCV13
  Arms: maternal group
Biological: placebo 0.9% sodium chloride plus tetanus toxoid — pregnant women will be given intramuscular saline injection between 28-34 weeks
  Other Names: placebo
  Arms: control group
Other: tetanus toxoid — new born babies will be given PCV13 vaccine at birth
  Arms: neonatal group

SUMMARY:
Streptococcus pneumoniae is responsible for over 10 percent of death in children under five and many of these deaths occur in early infancy before the current pneumococcal schedule is effective and nearly half occur in sub Saharan Africa.

The PROPEL trial will examine the effect of either a maternal or a neonatal dose of a pneumococcal conjugate vaccine on pneumococcal colonisation in the nose which can be used to measure the risk of disease in early life.

600 Expectant mothers will be randomized at between 28 and 34 weeks to a maternal group, a neonatal group or a control group in equal number (200 per group). Their subsequent born offspring will be followed up until nine months of age. Infants born from expectant mothers in the maternal and control group will receive their subsequent pneumococcal conjugate vaccination according to the national Expanded Programme on Immunisation (EPI) schedule in the Gambia at 8, 12 and 16 weeks while infants born to expectant mothers in the control group will receive the pneumococcal conjugate vaccine within 48 hours of birth and at 8 and 16 weeks of life. Randomization will be undertaken by defined un-blinded members of the clinical trial team who will be delegated for this task and who will not be involved in any other trial related procedures Pregnant women who are willing and who are identified by the staff of the government antenatal clinic as being potentially eligible according to gestation (assessed initially according to the date of the last menstrual period (LMP) - if known, or the fundal height), will be referred to a member of the clinical trial team.

Those who remain interested in participation having had the details of the study explained will have basic demographic, obstetric and contact details collected and will be invited, at a time of their convenience, to the Medical Research Council (MRC) clinical trial site for the formal informed consent process to be completed. Following informed consent, pregnancy will be confirmed with a urinary pregnancy test. Initial screening (e.g. for past-obstetric history and past-medical history etc) will be undertaken at this point along with screening bloods for serology (HIV, hepatitis B and syphilis) and haematology (haemoglobin and sickle test). A dating ultrasound scan (USS) will also be undertaken by designated clinical trial staff. On completion of screening, expectant mothers who are confirmed to be eligible according to the defined inclusion and exclusion criteria will be enrolled and randomized in parallel into one of three equally sized groups mentioned above (maternal, neonatal, control).

According to the group into which they have been randomized, mothers will receive a dose of PCV13 and tetanus toxoid [maternal group], placebo (0.9% sodium chloride) and tetanus toxoid [control group] or tetanus toxoid alone [neonatal group]. From this point on, the maternal and control groups (now 'Routine EPI Schedule') will be followed up in exactly the same way for the purposes of interventions and all endpoint assessments. Infants in the neonatal group ('Neonatal Schedule') will be followed up according to the schedule outlined.

At the time of presentation to the delivery unit a blood sample for serology and malaria Rapid Diagnostic Test (RDT) and an nasopharyngeal swab (NPS) sample will be obtained prior to or shortly following delivery. Immediately following delivery a sample of cord blood will be obtained and as soon as possible an NPS sample will be taken from the newborn. Anthropometric measurements will be taken from the newborn and an examination conducted. Once there has not been any contraindication to vaccination identified, all newborns will be administered the routine EPI vaccines according to the schedule in The Gambia (BCG, Hepatitis B and OPV). Those newborns in the Neonatal group will additionally be administered a single intramuscular (IM) dose of PCV13. At two, three and four months, infants will be administered the routine EPI vaccines. Those infants in the Maternal and Control Groups (Routine EPI Schedule) will additionally receive PCV13 at eight, 12, and 16 weeks while those in the Neonatal group will receive the vaccine at eight and 16 weeks only having received the first dose at birth. All infants will additionally receive a single dose of the inactivated poliovirus vaccine (IPV) at 16 weeks in line with the routine EPI schedule in The Gambia.

Following the vaccines administered to expectant mothers and following the vaccines administered at birth, home visits will be undertaken on day 1 to 6 to collect solicited local and systemic adverse (for PCV only) reactions and any unsolicited. A day 7 safety clinic visit will be conducted following the vaccines administered to expectant mothers and following the vaccines administered at birth. Infant will attend the clinical trial site for NPS and blood samples to be taken at specific time points.

DETAILED DESCRIPTION:
Members of the clinical trial team will base themselves within the government run antenatal clinics at the clinical trial sites in order to identify potentially eligible pregnant women. Working closely alongside government midwifery and nursing staff they will aim to identify pregnant women who are yet to reach 34 weeks gestation and who are thus potentially eligible for enrolment. Assessment of gestation at this first contact point will be based on the date of the LMP or the assessment of fundal height as is local practice (gestational age will be confirmed by ultrasound scanning once informed consent has been obtained and ultrasound based assessment will be used to determine final eligibility).

A member of the clinical trial team will discuss the study with potentially eligible expectant mothers who are provisionally interested and agree to receive this additional information. The discussion will be based on the contents of the informed consent document (ICD) and a copy of the ICD will be provided to the expectant mother at the end of the discussion.

Potentially eligible women who are interested will be encouraged to discuss the study with their spouse and other family members as appropriate. Following individual sensitization of the mother, a member of the field team may provide information to other family members (particularly the spouse) either by telephone or through a visit to the subject's residence according to the preference of the mother.

Expectant mothers who express an interest in participation will then be contacted to arrange a visit to the clinical trial site where informed consent will be undertaken. Written/thumb-printed informed consent will only be required from the expectant mother but in all cases it will be confirmed directly with the spouse (the father of the unborn baby) that they are aware of the study and have given their agreement. In the case of expectant mothers who are literate in English, they will be provided with a copy of the ICD but a member of the clinical trial team will nonetheless review the contents of the ICD line by line in English to ensure all details are covered and that the subject has the opportunity to ask questions regarding any aspect of the trial.

In the case of potential participants who are not literate in English but only in one of the local languages, a member of the clinical trial team fluent in the local language (as well as being English literate) will review the ICD line by line translating directly from the English ICD to the appropriate local language. In this case an impartial witness must be present throughout all elements of the consent process and must attest that the information on the ICD has been given accurately and in full. The impartial witness will also be required to sign the ICD to confirm that this has been the case.

Informed consent for study participation will be documented on the signature page of the ICD. The option to consent for the future use of any residual samples on study completion will also be given on the same page but the provision of such additional consent is not required for participation in the main trial.

A certified copy of the ICD is provided to the participant unless it is refused for some reason in which case it will be filed at the trial site. Such refusal must be documented in the subject's file so it is clear that the subject has been offered a copy The study will randomize 600 pregnant women at between 28 and 34 weeks gestation. Mothers will not be replaced following randomization. Screening of potentially eligible women will continue until this number is reached unless the trial is stopped for some other reason.

No further selection or assessment of eligibility will be undertaken on the newborn infants. All data will be included in the safety reporting irrespective of pregnancy outcome and safety follow-up should occur as planned for all infants. An infant may be excluded from the trial for the purposes of vaccination and/or clinical sampling if ongoing participation is considered to be against their best interests or if a contraindication to vaccination and/or to the obtaining of clinical samples is identified. An infant excluded in this way would not be replaced and hence this would not alter the target sample size of 600 pregnant women.

ELIGIBILITY:
Inclusion Criteria:

* Signed/thumb-printed informed consent for trial participation obtained*
* Pregnant woman aged between 18 and 40 years of age inclusive10*
* Singleton pregnancy*
* From 28 to 34 weeks11 gestation as determined by USS
* Resident within easy reach of the clinical trial site (no fixed boundaries will be set and such judgements will be made on a case by case basis by members of the field team in discussion with the potential participant, taking into account knowledge of the local transport links and geography)*
* Intention to deliver at the health centre related to the clinical trial site (i.e. Sukuta and Faji Kunda health centres)*
* Willingness and capacity to comply with all the study procedures, including those relating to the newborn infant, in the opinion of the principal investigator or designee

Exclusion Criteria:

* History of pre-eclampsia or eclampsia
* History of gestational diabetes
* Previous late stillbirth (defined as loss of pregnancy at any time after 28 weeks gestation)
* Previous premature delivery (defined as delivery before 37 weeks gestation)
* Previous neonatal death (defined as death of an infant within the first 28 days of life)
* Previous Caesarean section
* Previous delivery of an infant with major congenital anomalies
* Previous delivery of an infant with a known or suspected genetic or chromosomal abnormality
* History of other significant pregnancy related complications judged likely to affect the safety of the mother or infant or to significantly compromise the endpoint data collected
* History of other significant neonatal complications judged likely to affect the safety of the mother or infant or to significantly compromise the endpoint data collected
* Significant complications in current pregnancy
* Significant alcohol consumption during current pregnancy
* Significant maternal chronic illness including but not limited to hypertension requiring treatment, heart disease, lung disease, neurological disorders including a history of epilepsy or recurrent afebrile seizures, kidney disease, liver disease, anaemia and other haematological disorders, endocrine disorders including known diabetes mellitus, autoimmunity
* Severe anaemia (<7.0g/dL)[51]
* Known Human Immunodeficiency Virus (HIV) or hepatitis B (HBV) virus positive or found to be HIV or HBV positive during screening
* Positive result for syphilis infection on laboratory testing
* Known prior receipt of a pneumococcal vaccine (pneumococcal conjugate or pneumococcal polysaccharide vaccine)
* Receipt of any vaccine during the current pregnancy or plans to receive any non-study vaccines during the current pregnancy (tetanus toxoid vaccination is not an exclusion and vaccines given during national campaigns if applicable will not generally be exclusions)
* Any other condition judged to significantly increase the risks to either the mother or the infant within the current (including relevant history from previous pregnancies
* History of anaphylactic or severe allergic reactions to previous vaccines or history of anaphylactic or severe allergic reactions in previous offspring (if applicable)
* Receipt of any blood product including human immunoglobulins at any stage during the current pregnancy or plan to receive any blood products during the period or trial participation (receipt or blood products in an emergency or for obstetric reasons will not represent a protocol deviation given such situations are unplanned)
* Receipt of immunosuppressive or immuno-modulatory medication at any stage during the current pregnancy or plan to receive any such medication during the period or trial participation
* Clinically suspected or confirmed congenital or acquired clotting or bleeding disorders or the current receipt of medications known to alter clotting or bleeding
* Current malaria infection (on the day of randomization and vaccination)
* Any clinically significant signs or symptoms of acute illness, significant abnormalities in vital signs, an axillary temperature of > 37.5°C or any recorded fever (> 37.5°C) in the preceding 24 hours.
* 2 or more symptoms (nausea/vomiting, diarrhoea, headaches, fatigue and myalgia) rated as grade 2 and clinically significant on the maternal systemic reactogenicity scale present at baseline on the day of vaccination

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 600 (Estimated)
Dates: Start 2016-03-11 (Actual); Primary Completion 2019-02-19 (Actual); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
safety in pregnant mothers (SAE) | from 28 weeks gestation to 8 weeks after delivery
  SAE in expectant mothers from enrollment at 28 to 34 weeks gestation up to eight weeks from the end of the pregnancy
safety in newborns (SAE) | from birth until nine months of age
  SAE in infants from birth until nine months of age
safety in vaccinated pregnant women (local and systemic reactogenicity) | within the first seven days from vaccination
  Local and systemic reactogenicity within the first seven days of PCV13 administration to expectant mothers at between 28 and 34 weeks gestation
safety in vaccinated newborns (local and systemic reactogenicity) | within the first seven days from vaccination
  Local and systemic reactogenicity within the first seven days of PCV13 administration to newborn infants within the first week of life
outcome of pregnancy | from 28 weeks of gestation to delivery
  Pregnancy outcome
cumulative carriage acquisition rate in infants | from birth to 20 weeks of age
  collection of Naso Pharyngeal Swab to assess Vaccine Type (VT) pneumococcal carriage rate

SECONDARY OUTCOMES:
pneumococcal nasopharyngeal carriage rate of pregnant women | at delivery and at 8 weeks after delivery
  Nasopharyngeal carriage rate of total and VT pneumococcus in the mothers at delivery and at eight weeks following delivery
nasopharyngeal carriage rate of infants | form birth up to nine months of age
  Nasopharyngeal carriage rate of total and VT pneumococcus in infants up to nine months of age
pneumococcal vaccine type specific Immunoglobulin G (IgG) Geometric Mean Concentration (GMC) and sero protection rates in mothers and infants | at delivery and 8 weeks post delivery for the mothers and for the infants at birth, 8 weeks, 20 weeks and 9 months
  quantitative antibodies measurements and sero protection rate for both mothers and infants
opsonophagocytic antibodies titres in infants | at birth, 8 & 20 weeks of age
  qualitative antibodies measurements in infants
polio virus type 1,2,3, Geometric Mean Titre (GMT) and hepatitis B GMC sero protection rate in infants | at 8 weeks of age
  effect of co-administration of PCV13 with polio and hepatitis B vaccines
diptheria toxoid GMC sero protection rate | at birth, 8 & 20 weeks of age
  the effect of the diptheria mutant carrier protein on subsequent vaccination to the infants
tetanus toxoid GMC sero protection rate in mothers | at birth
  effect of co-administration with PCV13

CONTACTS AND LOCATIONS:
Overall Officials: Ed Clarke, MB, Principal Investigator — Medical Research Council Unit, The Gambia
Locations (1):
- Sukuta Health Centre, Banjul, The Gambia